CLINICAL TRIAL: NCT07257029
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled Trial of Topical Ketotifen Fumarate 0.25% Cream for Females With Secondary Vestibulodynia
Brief Title: Topical Ketotifen 0.25% for Secondary Vestibulodynia
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Center for Vulvovaginal Disorders (Other)
Collaborators: National Vulvodynia Association (Other)
Responsible Party: Principal Investigator, Andrew T. Goldstein, MD, Medical Director, Center for Vulvovaginal Disorders, Center for Vulvovaginal Disorders
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CVVD-KF1
Record Dates: First submitted 2025-11-21; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Provoked Vestibulodynia; Secondary Provoked Vestibulodynia; Vulvodynia; Vulvary Pain Disorders; Neuroproliferative Vestibulodynia; Mast Cell-mediated Neuroinflammation; Instertional Dyspareunia
Keywords: ketotifen fumarate; vulvodynia; provoked vestibulodynia; secondary vestibulodynia; vulvar pain; insertional dyspareunia; mast cell stabilizer; neuroproliferative pain; topical antihistamine; vulvar vestibule; non-hormonal treatment; vestibular tenderness; female sexual pain; vestibulodynia clinical trial; vulvar pain disorder; randomized controlled trial; algometer; dilator test; vulvodynia experience questionnaire (VEQ)
MeSH Terms: conditions — Vulvodynia | interventions — Ketotifen

STUDY DESIGN:
Intervention Model Description: This is a multi-center, randomized, double-blind, placebo-controlled, parallel-assignment Phase 2 trial. After a 2-week single-blind placebo run-in, eligible participants are randomized 1:1 to receive topical ketotifen fumarate 0.25% cream or matching vehicle cream. Participants apply their assigned treatment twice daily for 12 weeks, with no crossover between study arms. All investigators, participants, and study staff remain blinded to assignment until database lock.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ketotifen Fumarate 0.25% Cream (Experimental): Participants receive topical ketotifen fumarate 0.25% cream applied as a thin layer to the vulvar vestibule twice daily (approximately every 8-12 hours) for 12 weeks following completion of the 2-week placebo run-in period. The ketotifen cream is supplied in pre-weighed tubes and used for the full randomized treatment phase.
  Interventions: Drug: Ketotifen Fumarate 0.25% Cream
- Placebo (Vehicle Cream) (Placebo Comparator): Participants receive the matching vehicle cream applied as a thin layer to the vulvar vestibule twice daily (approximately every 8-12 hours) for 12 weeks following completion of the 2-week placebo run-in period. The placebo cream is identical in appearance and packaging to the active study cream and is supplied in pre-weighed tubes for the full randomized treatment phase.
  Interventions: Drug: Placebo (Vehicle Cream)

INTERVENTIONS:
Drug: Ketotifen Fumarate 0.25% Cream — Participants apply topical ketotifen fumarate 0.25% cream as a thin layer to the vulvar vestibule twice daily (approximately every 8-12 hours) for 12 weeks after completing the 2-week placebo run-in period. The cream is provided in pre-weighed tubes and used throughout the randomized treatment phase.
  Arms: Ketotifen Fumarate 0.25% Cream
Drug: Placebo (Vehicle Cream) — Participants apply the matching vehicle cream as a thin layer to the vulvar vestibule twice daily (approximately every 8-12 hours) for 12 weeks following completion of the 2-week placebo run-in period. The placebo cream is identical in appearance and packaging to the ketotifen cream and is provided in pre-weighed tubes for use throughout the randomized treatment phase.
  Arms: Placebo (Vehicle Cream)

SUMMARY:
This is a Phase 2, multi-center, randomized, double-blind, placebo-controlled trial evaluating the safety and efficacy of topical ketotifen fumarate 0.25% cream in adult women with secondary provoked vestibulodynia (PVD). Secondary PVD is a chronic vulvar pain condition characterized by burning or sharp pain with vaginal penetration (e.g., intercourse, tampon use) and touch of the vulvar vestibule, often following recurrent infections or topical irritant exposures. Preclinical studies suggest that ketotifen, a mast-cell stabilizer and histamine H1 antagonist, may reduce neuroinflammation and abnormal nerve growth in the vulvar vestibule, offering a mechanism-based, non-surgical treatment option.

Approximately 54 women aged 18 years and older who meet ISSVD/ISSWSH/IPPS criteria for secondary PVD without vulvovaginal atrophy will be enrolled. After a 1-week screening period, all participants will complete a 2-week single-blind placebo run-in; those with a strong placebo response or intolerance to vehicle cream will not be randomized. Eligible participants will then be randomized 1:1 to receive ketotifen fumarate 0.25% cream or matching placebo cream applied twice daily to the vulvar vestibule for 12 weeks.

The primary outcome is change from baseline to Week 15 in pain intensity with the baseline dilator maximum tested size (DMTS), measured on an 11-point numeric rating scale. Secondary outcomes include changes in Vulvodynia Experience Questionnaire (VEQ) scores, vestibular pain thresholds measured by Wagner algometry, and participant-reported meaningful benefit at the end of treatment. Safety assessments will include adverse events, application-site reactions, physical examinations, vital signs, and pregnancy testing. This study will provide the first controlled clinical data on topical ketotifen for secondary PVD and inform the feasibility of larger registration trials.

DETAILED DESCRIPTION:
This Phase 2 clinical trial is designed to evaluate a novel, mechanism-based topical treatment for secondary provoked vestibulodynia (PVD), a chronic pain condition affecting the vulvar vestibule. Women with PVD commonly describe burning, stinging, or sharp pain with tampon insertion, penetrative sexual activity, or light touch to the vestibular tissue. Many have lived with symptoms for years, and the condition can severely impair sexual function, intimate relationships, and overall quality of life. At present, there are no FDA-approved pharmacologic options, and the most effective intervention, vestibulectomy (surgical excision of painful vestibular tissue), is invasive and often unacceptable to patients.

Histopathologic and translational research has begun to clarify biological mechanisms that may drive PVD, particularly in women whose symptoms arise after recurrent vulvovaginal candidiasis or exposure to topical irritants. Vestibular tissue samples from patients undergoing vestibulectomy consistently show increased nerve density and clusters of activated mast cells within the mucosa. These findings support a model in which recurrent or persistent inflammation leads to mast-cell activation, release of pro-inflammatory mediators (including histamine and nerve growth factor), and pathologic neuroproliferation in the vestibular tissue. Preclinical work in rodent models has further demonstrated that repeated vulvovaginal fungal infections can induce chronic vulvar pain, even after clearance of infection, and that mast cell-derived factors are key contributors to sustained hypersensitivity and abnormal innervation.

Ketotifen fumarate is an oral and topical antihistamine with dual activity as a non-competitive H1 receptor antagonist and mast-cell stabilizer. It has decades of clinical use in allergic disorders and asthma prophylaxis and is generally well tolerated when used chronically. In a validated rat model mimicking PVD, ketotifen reduced vulvar mechanical and thermal hypersensitivity, decreased mast-cell activation and accumulation, lowered levels of nerve growth factor, and limited excessive nerve fiber growth in the vestibule. Modulation of these neuroinflammatory pathways suggests that ketotifen may attenuate the central biological processes driving pain in secondary PVD.

On the basis of this mechanistic rationale, an international vulvodynia summit of clinicians, scientists, and patient stakeholders recently reviewed potential candidates for future clinical trials in PVD. Ketotifen emerged as the highest-priority medication to move forward into human studies for neuroproliferative, inflammation-driven PVD. However, to date, no randomized, placebo-controlled clinical trial has tested topical ketotifen for this indication. This trial is designed to fill that gap by rigorously evaluating efficacy, safety, and tolerability of a 0.25% ketotifen fumarate cream applied directly to the vulvar vestibule.

Study Objectives

The overarching goal of the study is to determine whether topical ketotifen fumarate 0.25% cream improves pain and function in women with secondary PVD, compared with a matching vehicle cream. Specific aims are:

Efficacy:

To determine whether 12 weeks of twice-daily topical ketotifen reduces pain with vaginal dilator insertion at a standardized, participant-specific dilator size, as measured by an 11-point numeric rating scale (NRS).

To explore whether ketotifen improves broader domains of PVD-related symptoms and functioning, including daily pain, sexual function, and quality of life, using a validated vulvodynia-specific patient-reported outcome measure.

To assess changes in objective vestibular pain thresholds using standardized pressure algometry.

Safety and Tolerability:

To characterize local tolerability at the application site (e.g., burning, stinging, pruritus, erythema) with topical ketotifen versus vehicle.

To monitor for systemic adverse events potentially related to antihistaminic or anticholinergic activity, although systemic absorption is expected to be minimal with localized application.

Feasibility:

To determine feasibility of recruitment, completion of the placebo run-in, adherence to a twice-daily application regimen over 12 weeks, and retention through the Week 15 endpoint in a multi-center setting dedicated to vulvovaginal disorders.

To evaluate whether a placebo run-in enriches the randomized sample by excluding strong placebo responders and participants intolerant of the vehicle cream.

Study Design and Setting This is a multi-center, randomized, double-blind, vehicle-controlled Phase 2 study conducted at three specialized vulvovaginal disorders centers in the United States (New York, Washington, DC, and Tampa, Florida). Participants are adult women (≥18 years) with a clinical diagnosis of secondary provoked vestibulodynia, defined by consensus criteria from ISSVD/ISSWSH/IPPS and characterized by localized vestibular tenderness with associated inflammatory and neuroproliferative features, in the absence of vulvovaginal atrophy.

Each participant's involvement spans approximately 15 weeks, including:

Screening period (up to 1 week prior to placebo initiation): confirmation of eligibility, review of medical and vulvar pain history, physical and gynecologic examination, vaginal cultures to rule out infection, baseline pain and functional assessments, and pregnancy testing where applicable.

Single-blind placebo run-in (2 weeks): all eligible participants apply vehicle cream twice daily to the vulvar vestibule. This phase is designed to identify individuals who either respond substantially to vehicle alone or cannot tolerate the cream base.

Randomized double-blind treatment (12 weeks): participants who remain eligible and do not meet run-in exclusion criteria are randomized 1:1 to receive topical ketotifen fumarate 0.25% cream or vehicle, applied twice daily to the affected vestibular area(s).

Study visits are scheduled at Screening (Day 0), Week 3 (randomization visit), Week 9 (mid-treatment assessment), and Week 15 (end-of-treatment assessment). A safety follow-up period of 30 days after the last application of study treatment is planned, during which adverse events can still be reported.

To accommodate real-world scheduling challenges, visits are allowed within protocol-specified time windows. Minor deviations within a limited window will be recorded but do not necessarily exclude participants from the per-protocol analysis, whereas more substantial delays may be classified as major protocol deviations and can lead to exclusion from the per-protocol population at the investigators' discretion.

Interventions Participants will apply a thin layer of study cream (ketotifen fumarate 0.25% or vehicle) to the vulvar vestibule twice daily, approximately 8-12 hours apart, for 12 consecutive weeks following the run-in. Application is intended to be directly over the painful vestibular sites identified at baseline, and participants are instructed not to apply the cream immediately before sexual activity.

Study drug is supplied in pre-weighed tubes. At each treatment visit, tubes are dispensed and collected to assess adherence via change in tube weight, complemented by participant self-report regarding missed doses or deviations in use. Drug accountability procedures ensure that only enrolled participants receive the investigational treatment and that temperature and storage conditions are monitored in accordance with product specifications.

Participants and all site personnel (investigators, staff, and outcome assessors) remain blinded to treatment assignment. Randomization is performed centrally by study staff using a secure randomization tool. Emergency unblinding is permitted only if knowledge of treatment assignment is judged essential for participant safety.

Concomitant medications are recorded from 30 days prior to first application of study cream through 30 days after the last application. Stable regimens for chronic medical conditions are allowed if not expected to interact with ketotifen's mechanism or study outcomes. Initiation or regimen changes in medications commonly used to treat chronic vulvar pain (e.g., gabapentinoids, tricyclic antidepressants, SSRIs/SNRIs, certain muscle relaxants), initiation of pelvic floor physical therapy, or introduction of new topical vulvar therapies are not permitted during the trial, in order to avoid confounding efficacy assessments.

Outcome Measures and Assessments The trial focuses on a clinically meaningful assessment of insertional pain and functional penetration capacity, supported by patient-reported outcome measures and quantitative sensory testing.

Primary Outcome The primary endpoint is the change from baseline to Week 15 in dilator-induced pain intensity at the participant's baseline dilator maximum tested size (DMTS), measured using an 11-point numeric rating scale (0 = no pain, 10 = worst imaginable pain).

At baseline and each follow-up visit, participants undergo a standardized vaginal dilator assessment with a graded set of dilators. The clinician determines the largest size that the participant can tolerate without unacceptable pain at baseline; this size is used as the reference for the primary pain outcome. This approach allows the study to evaluate whether ketotifen can reduce pain with a functionally relevant level of penetration, rather than only assessing tolerance of progressively larger dilators.

Key Secondary and Exploratory Outcomes

Dilator function and pain trajectory:

Changes in dilator-related pain and, where applicable, changes in DMTS size across visits are recorded to capture both symptomatic relief and possible improvements in functional capacity.

Vulvodynia Experience Questionnaire (VEQ):

A vulvodynia-specific, validated patient-reported outcome measure is administered at baseline, Week 3, Week 9, and Week 15. The VEQ assesses multiple domains relevant to PVD, including pain intensity, pain during sexual and non-sexual activities, emotional impact, and quality of life.

Vestibular pain thresholds (Wagner algometer):

Pressure pain thresholds are measured at six standardized vestibular sites using a handheld algometer that applies force at a fixed rate up to a predefined maximum. The force at which the participant first reports pain is recorded at each site, providing an objective measure of mechanical sensitivity.

Participant-perceived meaningful benefit:

At the end-of-treatment visit (Week 15), participants complete a brief questionnaire indicating whether they experienced a meaningful benefit from the study treatment. This patient-centered endpoint helps interpret the clinical relevance of changes in quantitative measures.

Safety and Tolerability

Safety assessments include:

Medical history and physical examinations at prespecified visits, with particular attention to the vulvar vestibule and surrounding tissue.

Vital signs at each in-person visit. Urine pregnancy tests for participants of childbearing potential at baseline and follow-up visits.

Continuous monitoring and documentation of adverse events (AEs) and serious adverse events (SAEs) from the time of consent through 30 days after the last study drug application.

Local application site events (e.g., burning, stinging, pruritus, erythema) are specifically elicited and recorded. Investigators grade severity according to CTCAE v5.0 and assess causality in relation to the study drug. Temporary interruption of treatment is permitted in the setting of intolerable local reactions or other concerning AEs; resumption may occur if symptoms improve and the investigator deems it safe. Permanent discontinuation is required for certain predefined scenarios, including persistent or severe intolerance or repeated vulvovaginal infections during the treatment window.

Study Population

The target population is adult women with a well-characterized, clinically confirmed diagnosis of secondary provoked vestibulodynia. Key elements include:

Age ≥18 years. Ability to read and understand English and to provide written informed consent. A history of at least 6 continuous months of insertional dyspareunia, pain with tampon insertion, or vestibular pain to light touch.

On physical examination, moderate to severe tenderness localized to the vulvar vestibule, consistent with secondary PVD and not attributable to vulvovaginal atrophy or other vulvar dermatoses.

Absence of active vulvovaginal infections at the time of randomization (infections discovered at screening can be treated and participants re-evaluated once cured).

Participants with significant surgery to the vestibule, active dermatoses, or concurrent painful vulvar conditions unrelated to PVD are excluded to reduce heterogeneity and avoid confounding. Medications and therapies that could significantly alter vestibular pain or interact with ketotifen's action are also restricted during the trial window. Women who are pregnant, breastfeeding, or unable to complete the dilator assessment at the smallest size during baseline evaluation are excluded.

The protocol does not exclude participation based on race or ethnicity, and recruitment is intended to reach a clinically diverse group of women seen at the participating specialty clinics.

Risk Mitigation and Partner Safety

Although systemic absorption of topical ketotifen applied to the vulvar vestibule is expected to be low, several precautions are built into the protocol:

Participants are counseled to use barrier protection (e.g., male condoms) during vaginal intercourse throughout the study to minimize the possibility of partner exposure to the investigational product.

Participants are instructed to refrain from receiving oral sex to avoid direct ingestion of cream by partners.

New topical agents or over-the-counter vulvar creams are discouraged unless approved by the investigator, to minimize irritant or allergic reactions and avoid confounding safety assessments.

Participants are closely monitored for signs of local irritation and for systemic effects potentially attributable to antihistaminic or anticholinergic activity (such as sedation, dizziness, or dry mouth), though these are considered unlikely with the topical route and concentration used.

Statistical Considerations The sample size was determined to provide adequate power to detect a clinically meaningful difference in the primary pain outcome between ketotifen and vehicle. Assuming a response rate of 25% in the placebo group and 65% in the active treatment group, a total of 48 completers (24 per arm) yields approximately 80% power at a two-sided alpha of 0.05. Allowing for an anticipated dropout rate of about 10%, the study aims to randomize 54 participants (27 per arm). Participants who drop out or are withdrawn after randomization will remain in the intent-to-treat analyses when possible.

The primary analysis will be conducted in the intent-to-treat population using a repeated-measures model that incorporates treatment group, visit, treatment-by-visit interaction, and study site as fixed effects, with baseline pain at the reference dilator size as a covariate. Least-squares mean differences between treatment groups at Week 15 will be estimated with two-sided 95% confidence intervals. If model assumptions are not met, alternative rank-based or bootstrapped approaches will be employed as sensitivity analyses.

Secondary and exploratory outcomes, including VEQ scores, algometry thresholds, and meaningful benefit responses, will be analyzed using appropriate parametric or non-parametric methods. Given the exploratory nature of this Phase 2 trial, no formal multiplicity adjustment is planned. Safety analyses will summarize the incidence, severity, and relationship of AEs and SAEs across treatment groups.

Data Handling and Confidentiality Study data are captured in a secure, password-protected electronic database using de-identified participant codes. Source documents are maintained at the clinical sites in locked or access-restricted areas and may be inspected by regulatory authorities or oversight bodies in accordance with applicable regulations. Data quality assurance includes staff training, standardized procedures for key assessments (dilator testing, algometry, questionnaires), and periodic data reviews for completeness and internal consistency.

Potential Impact Secondary provoked vestibulodynia is a prevalent, under-recognized cause of chronic vulvar and sexual pain with limited evidence-based treatment options. Many affected women face years of trial-and-error therapies, substantial distress, and impaired quality of life. By targeting mast-cell-mediated neuroinflammation and abnormal innervation with a locally applied, non-hormonal agent that already has an established safety profile in other indications, this study seeks to provide the first controlled human data on topical ketotifen for PVD.

If the results demonstrate clinically meaningful improvements in pain and function with acceptable tolerability, the trial will lay the groundwork for larger, definitive registration studies. Ultimately, this line of research aims to expand the therapeutic toolkit for PVD beyond surgery and nonspecific off-label medications, moving toward mechanism-based, patient-centered, and less invasive treatment options for vulvar pain.

ELIGIBILITY:
Inclusion Criteria:

* Female participants ≥18 years of age
* Able to provide signed and dated informed consent
* Able to read, write, understand, and complete English-language study-related forms and communicate in English
* Has a stable address and is available for the duration of the study
* In good general health based on medical history
* Willing to comply with all study procedures
* Body mass index (BMI) between 18.5 kg/m² and 32.0 kg/m² (inclusive)
* Meets ISSVD/ISSWSH/IPPS criteria for secondary provoked vestibulodynia, including: 6 continuous months of vulvar symptoms (insertional dyspareunia, pain with tampon insertion, or pain to touch); moderate to severe vestibular tenderness to light touch on physical exam
* No evidence of vulvovaginal atrophy
* If atrophy is present, must complete ≥12 weeks of topical hormone therapy and be re-screened to confirm resolution before enrollment
* Negative vaginal culture for infection at randomization (participants with positive cultures at screening may be treated and retested)

Exclusion Criteria:

* Pregnancy or lactation
* Unable to tolerate the smallest dilator during baseline dilator assessment
* Active vaginal infection (Candida, BV, trichomonas, HSV)
* May re-screen after treatment and documented cure
* Active cutaneous disease of the vestibule
* Current presentation of other painful vulvar conditions, including:

Pudendal neuralgia Lichen sclerosus Lichen planus Plasma cell vulvitis Vulvar intraepithelial neoplasia Sjögren's disease Desquamative inflammatory vaginitis

* Hypoestrogenic states (e.g., vulvar atrophy due to menopause or medications)
* History of significant vestibular or vaginal surgery, including:

Vestibulectomy Perineoplasty Bladder neck suspension Anterior/posterior colporrhaphy Pudendal nerve neurolysis Ablative or fractional laser procedures

* Initiation or planned change in any of the following within 30 days before screening or during the study:

Gabapentinoids Tricyclic antidepressants SSRIs or SNRIs Hormone replacement therapy Systemic or local muscle relaxants (benzodiazepines, baclofen, botulinum toxin, cyclobenzaprine, CBD suppositories) Pelvic floor physical therapy

* Use of another investigational drug or intervention within the past 3 months
* Positive vaginal culture during the study requiring two or more treatments (per protocol, second infection leads to termination)
* Any condition or factor that, in the opinion of the investigator, would interfere with study participation or safety

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2026-01-02 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in Dilator-Induced Pain at the Baseline Dilator Maximum Tested Size (DMTS) | Baseline to Week 15
  Pain intensity is measured using the 11-point Numeric Rating Scale (0-10) at the participant's baseline dilator maximum tested size during standardized dilator testing. This assesses change in insertional pain from baseline over the randomized treatment period.

SECONDARY OUTCOMES:
Change in Vulvodynia Experience Questionnaire (VEQ) Scores | Baseline, Week 3, Week 9, Week 15.
  Change from baseline in patient-reported symptoms, function, and quality of life using the validated VEQ instrument administered at each study visit.
Change in Vestibular Pain Thresholds (Wagner Algometer) | Baseline, Week 3, Week 9, Week 15.
  Mechanical pain thresholds measured at six standardized vestibular sites using a Wagner algometer applying force at 0.5 N/s. Threshold recorded when the participant first reports pain.
Patient-Reported Meaningful Benefit | Week 15
  Participant-reported global assessment asking whether the treatment provided meaningful benefit.

OTHER OUTCOMES:
Incidence of Adverse Events (AEs) | From first application through 30 days after last dose
  Frequency and type of treatment-emergency adverse events
Incidence of Serious Adverse Events (SAEs) | From informed consent through 30 days after last dose
  Number of serious adverse events meeting regulatory criteria
Local Application Site Reactions | Baseline, Week 3, Week 9, Week 15
  Incidence of stinging, burning, pruritis, erythema, or related reactions at applications site

CONTACTS AND LOCATIONS:
Overall Officials: Andrew T Goldstein, MD, Principal Investigator — Center for Vulvovaginal Disorders
Locations (3):
- United States (3):
  - The Center for Vulvovaginal Disorders - Washington, DC, Washington D.C., District of Columbia
  - The Center for Vulvovaginal Disorders, Tampa, Florida
  - The Center for Vulvovaginal Disorders - New York, New York, New York

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared. The study database will not be made publicly available due to privacy considerations and lack of a formal data-sharing plan.

REFERENCES:
- [Background] Tympanidis P, Terenghi G, Dowd P. Increased innervation of the vulval vestibule in patients with vulvodynia. Br J Dermatol. 2003 May;148(5):1021-7. doi: 10.1046/j.1365-2133.2003.05308.x. PMID 12786836
- [Background] Gagnon C, Minton J, Goldstein I. Vestibular anesthesia test for neuroproliferative vestibulodynia. J Sex Med. 2014 Aug;11(8):1888-91. doi: 10.1111/jsm.12630. No abstract available. PMID 25066059
- [Background] Goldstein AT, Pukall CF, Brown C, Bergeron S, Stein A, Kellogg-Spadt S. Vulvodynia: Assessment and Treatment. J Sex Med. 2016 Apr;13(4):572-90. doi: 10.1016/j.jsxm.2016.01.020. Epub 2016 Mar 25. PMID 27045258
- [Background] Awad-Igbaria Y, Edelman D, Ianshin E, Abu-Ata S, Shamir A, Bornstein J, Palzur E. Inflammation-induced mast cell-derived nerve growth factor: a key player in chronic vulvar pain? Brain. 2025 Jan 7;148(1):331-346. doi: 10.1093/brain/awae228. PMID 39001871
- [Background] Awad-Igbaria Y, Dadon S, Shamir A, Livoff A, Shlapobersky M, Bornstein J, Palzur E. Characterization of Early Inflammatory Events Leading to Provoked Vulvodynia Development in Rats. J Inflamm Res. 2022 Jul 11;15:3901-3923. doi: 10.2147/JIR.S367193. eCollection 2022. PMID 35845089
- [Background] Drian A, Goldstein SW, Kim NN, Goldstein AS, Hartzell-Cushanick R, Yee A, Goldstein I. Immunohistochemical staining with CD117 and PGP9.5 of excised vestibular tissue from patients with neuroproliferative vestibulodynia. J Sex Med. 2024 Apr 30;21(5):479-493. doi: 10.1093/jsxmed/qdae030. PMID 38521973
- [Background] Bornstein J, Bogliatto F, Haefner HK, Stockdale CK, Preti M, Bohl TG, Reutter J; ISSVD Terminology Committee. The 2015 International Society for the Study of Vulvovaginal Disease (ISSVD) Terminology of Vulvar Squamous Intraepithelial Lesions. Obstet Gynecol. 2016 Feb;127(2):264-8. doi: 10.1097/AOG.0000000000001285. PMID 26942352